CLINICAL TRIAL: NCT05175872
Title: Factors Affecting Mortality and Morbidity in Trauma Patients Followed in Intensive Care Unit
Acronym: trauma
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Cansu Kilinc Berktas, Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 928
Record Dates: First submitted 2020-01-03; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Trauma, Multiple; Trauma Injury
Keywords: trauma; mortality; morbidity
MeSH Terms: conditions — Multiple Trauma; Accidental Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the demographic and clinical characteristics of trauma patients followed up in the Intensive Care Unit of the Anesthesiology and Reanimation Clinic of the Health Sciences University Okmeydanı Training and Research Hospital for a 2-year period were evaluated prospectively to determine the morbidity and mortality rates and to determine the factors affecting these rates. data.

DETAILED DESCRIPTION:
Trauma is an important health problem that causes increased morbidity and mortality. Most of the patients are taken into intensive care and followed up in intensive care with severe and multitrauma and constitute an important part of the critical diseases followed in the intensive care unit. At the same time, these fatal injuries cause a serious public health problem both economically and socially.

According to World Health Organization data, 5.8 million people die each year due to trauma. Trauma is seen more frequently at a young age and the most common cause is motor vehicle accidents and it is the first cause of death between 1-44 years. There is a strong relationship between deaths caused by trauma and factors such as age, gender, cause of trauma, and trauma area. In addition, the duration of ICU and mechanical ventilator stay, supportive treatments, trauma scores, and scores such as APACHE 2 and SOFA routinely used in intensive care have been shown to be strongly associated with mortality.

Therefore, the demographic data, trauma scores, mechanical ventilator requirement, renal failure, inotropic need, intensive care scores such as APACHE 2, SOFA, re-operation, re-operation, intensive care stay, blood replacement need, wound infection and morbidity and mortality in trauma patients will be effective.

ELIGIBILITY:
Inclusion Criteria:

* Trauma Patients Followed up in the Intensive Care Unit between 14 October 2019 and 15 October 2021
* All trauma patients over the age of 18 who signed the informed consent form and agreed to participate in the trial

Exclusion Criteria:

* Patients under the age of 18
* Patients who refused to participate in the study
* Non-traumatic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All trauma patients older than 18 years of age followed up in the anesthesia and reanimation unit of the investigator's hospital with the approval of the Ethics Committee of Okmeydanı Training and Research Hospital will be included in the study.
Sampling Method: Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Injury Severity Score | during the procedure
  The Injury Severity Score (ISS) assesses the combined effects of the multiply-injured patients and is based on an anatomical injury severity classification.
  The ISS is calculated as the sum of the squares of the highest AIS code in each of the three most severely injured ISS body regions. These body regions are:
  * Head or neck
  * Face
  * Chest
  * Abdominal or pelvic contents
  * Extremities or pelvic girdle
  * External Injury Severity Scores range from 1 to 75. If an injury is assigned an AIS of 6 (identifying a currently untreatable injury), the ISS score is automatically assigned 75.
Clinical features | during the procedure
  Inotropic requirement, renal failure, mechanical ventilation requirement, re-operation, need for intensive care unit, blood replacement requirement, wound infection, discharge from intensive care unit, 28-day mortality, hospital mortality, mortality, number of stay days in intensive care unit during intensive care follow-up , 20/5000 history of drug use and hospital stay days will be recorded.

SECONDARY OUTCOMES:
Surgical Apgar Score | during the procedure
  Surgical Apgar Score (SAS) is used for predicting the occurrence of major postoperative morbidities and mortality after general and vascular surgery. SAS is a 10-point score based on 3 easily obtained parameters: the estimated blood loss, lowest heart rate, and lowest mean arterial pressure during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Namigar Turgut, Prof.Dr., Study Director — Okmeydani Education and Research Hospital
Locations (1):
- Okmeydani Education and Research Hospital, Istanbul, Turkey (Türkiye)